CLINICAL TRIAL: NCT01388465
Title: Feasibility of Using Text-Message Support to Improve Antibiotic Adherence After ED Discharge
Brief Title: Text-message Support to Improve Oral Antibiotic Adherence After ED Discharge
Acronym: ImpACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO11020492
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Medication Adherence
Keywords: Adherence; Intervention
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile phone text message Intervention (Experimental): Daily assessments with feedback about (1) filling prescription and (2) number of doses taken
  Interventions: Behavioral: Mobile phone text messaging
- Control (No Intervention): No TM queries or feedback

INTERVENTIONS:
Behavioral: Mobile phone text messaging — Daily assessment followed by feedback
  Arms: Mobile phone text message Intervention

SUMMARY:
The investigators are testing the hypothesis that patients who are exposed to daily text-message (TM) assessments with feedback will have better adherence to prescription than those patients not exposed to TM-based queries with feedback.

DETAILED DESCRIPTION:
Short course, oral antibiotics are frequently prescribed to patients treated/discharged from the Emergency Department. Medication adherence involves the patient taking the proper daily dosing of prescribed medication for the entire length of time it is prescribed. Previous studies have shown that prescription non-filling rates range from 5 to 20%. Other studies have shown that even if patients fill their prescription, as low as 30-40% will properly take the medication. The purpose of this study is to determine if the proportion of patients discharged from the Emergency Department that are adherent with antibiotics is higher in patients that are provided TM support using self-report.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Planned discharge form the ED on oral antibiotics

Exclusion Criteria:

* non-English speaking
* Prisoner
* No personal mobile phone with text message features

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Successfully picked up prescription within 24 hours of ED discharge | 24 hours post ED discharge
  We will compare the proporiton of participants in each group who have picked up their prescription within 24 hours of discharge

SECONDARY OUTCOMES:
Complete adherence to oral antibiotics | 3-14 days
  We will compare the proporiton of participants in either group who have achieved complete adherence to dosing and days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Mercy Emergency Department, Pittsburgh, Pennsylvania, United States